CLINICAL TRIAL: NCT05053503
Title: Delivering Transcutaneous Auricular Neurostimulation to Improve Relapse Prevention in Opioid Use Disorder
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Biomedical, Inc. (Industry)
Collaborators: Hazelden Betty Ford Foundation (Unknown); Gaudenzia, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SBM-OWP-03
Record Dates: First submitted 2021-08-16; First posted 2021-09-22 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Opioid-use Disorder; Opioid Withdrawal
Keywords: auricular neurostimulation; vagus nerve stimulation; transcutaneous; withdrawal symptoms; relapse prevention
MeSH Terms: conditions — Opioid-Related Disorders; Substance Withdrawal Syndrome | interventions — lofexidine

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled, multi-center, clinical trial in which participants with a history of dependence on prescriptive or non-prescriptive opioids will be randomized 2:1 into one of four treatment groups during Phase I (acute detoxification). Phase I will occur during the participant's treatment in a residential detox center. Participants will have the option to continue into Phase II of the trial at the conclusion of their stay in the residential detox treatment program. In Phase II, participants will be re-randomized 1:1 into one of two treatment groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study investigators will be blind to patient treatment group assignment. Furthermore, each clinical site will use qualified COWS assessors that will be blind to randomization group assignment. This will ensure a non-biased assessment of opioid withdrawal symptoms. Information regarding study intervention will be withheld from the blinded COWS assessors. All participants will be blinded to their group assignment during acute detox treatment (Phase I). Participants will not be unblinded to their Phase I treatment until study exit, which may occur at the end of Phase II for participants who continue in the study. Participants will not be blinded to their treatment group during Phase II.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Active tAN + placebo (Placebo Comparator): tAN will be delivered at a duty cycle of for 5 minutes ON and 10 seconds OFF for up to 168 hours (7 days) therapy duration. Stimulation intensity will be customized to the participants comfort level and within range of therapeutic effectiveness. Participants will receive 3 placebo pills four times per day for 7 days. The placebo will appear similar to lofexidine in size, shape, color, and smell to lofexidine.
  Interventions: Device: Sparrow Ascent Therapy System
- Active tAN + lofexidine (Active Comparator): tAN will be delivered at a duty cycle of for 5 minutes ON and 10 seconds OFF for up to 168 hours (7 days) therapy duration. Stimulation intensity will be customized to the participants comfort level and within range of therapeutic effectiveness. Participants will receive 3 lofexidine 0.18 mg/tablets four times per day (daily dose of 2.16 mg) for 7 days.
  Interventions: Device: Sparrow Ascent Therapy System; Drug: Lofexidine
- Sham tAN + placebo (No Intervention): Participants will have the earpiece applied and the cable connected to the Patient Controller, but tAN stimulation will not be turned on. Participants will receive 3 placebo pills four times per day for 7 days. The placebo will appear similar to lofexidine in size, shape, color, and smell to lofexidine.
- Sham tAN + lofexidine (Sham Comparator): Participants will have the earpiece applied and the cable connected to the Patient Controller, but tAN stimulation will not be turned on. Participants will receive 3 lofexidine 0.18 mg/tablets four times per day (daily dose of 2.16 mg) for 7 days.
  Interventions: Drug: Lofexidine
- extended-release injectable naltrexone (Active Comparator): Extended-release injectable naltrexone will be administered according to the clinical site's standard of care.
  Interventions: Drug: Extended-release injectable naltrexone
- Active tAN + extended-release injectable naltrexone (Experimental): Extended-release injectable naltrexone will be administered according to the clinical site's standard of care. Participants will be provided with a Spark Sparrow Ascent Therapy System and instructed to administer therapy according to the specified frequencies:
  * Month 1 (Days 1 - 28): a minimum of 2 hours per day at least 5 days a week
  * Month 2 (Days 29 - 56): a minimum of 2 hours per day at least 3 days a week
  * Month 3 (Days 57 - 90: a minimum of 2 hours per day at least 1 day per week
  Interventions: Device: Sparrow Ascent Therapy System; Drug: Extended-release injectable naltrexone

INTERVENTIONS:
Device: Sparrow Ascent Therapy System — Transcutaneous auricular neurostimulation (tAN)
  Arms: Active tAN + extended-release injectable naltrexone; Active tAN + lofexidine; Active tAN + placebo
Drug: Lofexidine — Participants will receive 3 lofexidine 0.18 mg/tablets four times per day (daily dose of 2.16 mg) for 7 days.
  Arms: Active tAN + lofexidine; Sham tAN + lofexidine
Drug: Extended-release injectable naltrexone — Participants will receive extended-release injectable naltrexone based on the clinical site's standard of care.
  Arms: Active tAN + extended-release injectable naltrexone; extended-release injectable naltrexone

SUMMARY:
The primary objective of this trial is to determine whether tAN can improve relapse prevention beyond that seen with extended-release injectable naltrexone during Phase II.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, multi-center, clinical trial in which participants with a history of dependence on prescriptive or non-prescriptive opioids will be randomized 2:1 into one of four treatment groups during Phase I (acute detoxification, 7 days):

1. Group 1: Active tAN + placebo
2. Group 2: Active tAN + lofexidine
3. Group 3: Sham tAN + placebo
4. Group 4: Sham tAN + lofexidine

Phase I will occur during the participant's treatment in a residential detox center. Participants will have the option to continue into Phase II of the trial at the conclusion of their stay in the residential detox treatment program. In Phase II, participants will be re-randomized 1:1 into one of two treatment groups and will return weekly for 90 days:

1. Group 1: Extended-release injectable naltrexone
2. Group 2: Active tAN + extended-release injectable naltrexone

ELIGIBILITY:
Inclusion Criteria

1. Participant shows signs of current opioid dependence; prescription or non-prescription
2. Participant COWS score is ≥ 8 or in the opinion of the investigator the participant is in mild to moderate withdrawal at the baseline assessment
3. Participant is between 18 and 65 years of age
4. Participant is English proficient
5. Participant is able to provide informed consent and function at an intellectual level sufficient for study requirements

Exclusion Criteria

1. Participant presents current evidence of an uncontrolled and/or clinically significant medical condition or psychiatric condition
2. Participant has a history of epileptic seizures
3. Participant has a history of neurological diseases or traumatic brain injury
4. Participants using long-acting opioids such as methadone or buprenorphine for a period of five or more consecutive days prior to enrollment
5. Participant has recent suicide attempt leading to current hospital admission or continued expressed suicidal ideation
6. Participant has presence of devices, e.g., pacemakers, cochlear prosthesis, neurostimulators
7. Participant has abnormal ear anatomy or ear infection present
8. Participant is unwilling to transition to opioid antagonist medication following acute detox treatment
9. Subject has significant current suicidal ideation within 30 days prior to Screening as evidenced by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) completed at Screening, that, in the opinion of the investigator, warrants exclusion from the trial
10. Women of childbearing potential, not using adequate contraception as per investigator judgment or not willing to comply with contraception for the duration of the study
11. Females who are pregnant or lactating
12. Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
14-Panel Urine Drug Screen | Weekly throughout Phase II (13 weeks)
  In Phase II, participants will provide a weekly urine sample to determine if opioids have been used in the past week (in conjunction with a self-report). A urine drug screen cup will be used to detect presence of: Amphetamines, Buprenorphine, Benzodiazepines, Cocaine, Ethyl Glucuronide, Fentanyl, Synthetic Marijuana, Ecstasy, Methamphetamines, Methadone, Opiates / Morphine, Oxycodone, Cannabinoid (Marijuana), and Tramadol. The urine drug screen cup also contains a temperature strip to confirm appropriate temperature of the sample and an adulteration panel for determination of sample tampering.
Self-Report of Drug Use | Weekly throughout Phase II (13 weeks)
  In Phase II, participants will be asked weekly to self-report any use of opioids to determine if opioids have been used in the past week (in conjunction with a UDS sample).

SECONDARY OUTCOMES:
Clinical Opiate Withdrawal Scale (COWS) | 60 minutes after treatment initiation (Day 1, Phase I)
  The Clinical Opiate Withdrawal Scale (COWS) is an 11-item scale designed to be administered by a clinician. This tool can be used in both inpatient and outpatient settings to reproducibly rate common signs and symptoms of opiate withdrawal and monitor these symptoms over time. The summed score for the complete scale can be used to help clinicians determine the stage or severity of opiate withdrawal and assess the level of physical dependence on opioids. Scores range between 0 and 48 where total score is the sum of all the items. A higher score indicates more severe withdrawal symptoms. Scores between 5 and 12 indicate mild withdrawal, scores between 13 and 24 indicate moderate withdrawal, scores between 25 and 36 indicate moderately severe withdrawal and scores greater than 36 indicate severe withdrawal. A COWS score reduction of 15% or greater for a given individual is considered clinically significant.
Short Opiate Withdrawal Scale-Gossop (SOWS-Gossop) | 60 minutes after treatment initiation (Day 1, Phase I)
  The SOWS-Gossop is an appropriate, precise, and sensitive measure to evaluate the symptoms of acute opioid withdrawal in research or clinical settings. The scale was derived from the original 32-item Opiate Withdrawal Scale to reduce redundancy while providing an equally sensitive measure of opioid withdrawal symptom severity appropriate for research and clinical practice. The assessment is a self-administered test used for the assessment of opiate withdrawal symptoms. The scale contains ten items: yawning, muscular tension, runny eyes, muscle twitching, pains, and aches, feeling of coldness, stomach cramps, insomnia, heart pounding, and feeling sick, making it easy and rapid to administer. The tool has a 4-point rating scale: 0 for 'none,' 1 for 'mild,' 2 for 'moderate,' and 3 for 'severe', with scores ranging from 0 to 30.
Clinical Opiate Withdrawal Scale (COWS) | 6 hours after treatment initiation (Day 1, Phase I)
  The Clinical Opiate Withdrawal Scale (COWS) is an 11-item scale designed to be administered by a clinician. This tool can be used in both inpatient and outpatient settings to reproducibly rate common signs and symptoms of opiate withdrawal and monitor these symptoms over time. The summed score for the complete scale can be used to help clinicians determine the stage or severity of opiate withdrawal and assess the level of physical dependence on opioids. Scores range between 0 and 48 where total score is the sum of all the items. A higher score indicates more severe withdrawal symptoms. Scores between 5 and 12 indicate mild withdrawal, scores between 13 and 24 indicate moderate withdrawal, scores between 25 and 36 indicate moderately severe withdrawal and scores greater than 36 indicate severe withdrawal. A COWS score reduction of 15% or greater for a given individual is considered clinically significant.
Short Opiate Withdrawal Scale-Gossop (SOWS-Gossop) | 6 hours after treatment initiation (Day 1, Phase I)
  The SOWS-Gossop is an appropriate, precise, and sensitive measure to evaluate the symptoms of acute opioid withdrawal in research or clinical settings. The scale was derived from the original 32-item Opiate Withdrawal Scale to reduce redundancy while providing an equally sensitive measure of opioid withdrawal symptom severity appropriate for research and clinical practice. The assessment is a self-administered test used for the assessment of opiate withdrawal symptoms. The scale contains ten items: yawning, muscular tension, runny eyes, muscle twitching, pains, and aches, feeling of coldness, stomach cramps, insomnia, heart pounding, and feeling sick, making it easy and rapid to administer. The tool has a 4-point rating scale: 0 for 'none,' 1 for 'mild,' 2 for 'moderate,' and 3 for 'severe', with scores ranging from 0 to 30.
Clinical Opiate Withdrawal Scale (COWS) | Daily on Days 2-7 of Phase I
  The Clinical Opiate Withdrawal Scale (COWS) is an 11-item scale designed to be administered by a clinician. This tool can be used in both inpatient and outpatient settings to reproducibly rate common signs and symptoms of opiate withdrawal and monitor these symptoms over time. The summed score for the complete scale can be used to help clinicians determine the stage or severity of opiate withdrawal and assess the level of physical dependence on opioids. Scores range between 0 and 48 where total score is the sum of all the items. A higher score indicates more severe withdrawal symptoms. Scores between 5 and 12 indicate mild withdrawal, scores between 13 and 24 indicate moderate withdrawal, scores between 25 and 36 indicate moderately severe withdrawal and scores greater than 36 indicate severe withdrawal. A COWS score reduction of 15% or greater for a given individual is considered clinically significant.
Short Opiate Withdrawal Scale-Gossop (SOWS-Gossop) | Daily on Days 2-7 of Phase I
  The SOWS-Gossop is an appropriate, precise, and sensitive measure to evaluate the symptoms of acute opioid withdrawal in research or clinical settings. The scale was derived from the original 32-item Opiate Withdrawal Scale to reduce redundancy while providing an equally sensitive measure of opioid withdrawal symptom severity appropriate for research and clinical practice. The assessment is a self-administered test used for the assessment of opiate withdrawal symptoms. The scale contains ten items: yawning, muscular tension, runny eyes, muscle twitching, pains, and aches, feeling of coldness, stomach cramps, insomnia, heart pounding, and feeling sick, making it easy and rapid to administer. The tool has a 4-point rating scale: 0 for 'none,' 1 for 'mild,' 2 for 'moderate,' and 3 for 'severe', with scores ranging from 0 to 30.
Opioid Craving Scale (OCS) | Weekly throughout Phase II (13 weeks)
  The 3-item Opioid Craving Scale was adapted from the 3-item Cocaine Craving Scale for use with opioids. The original 5-item version was found to be valid and unidimensional among cocaine-dependent individuals. Participants are asked to answer the following three questions with responses ranging from 0-10, where 0 = Not at all and 10 = Extremely. Total possible score ranges from 0 to 30 with greater scores indicating higher opioid craving.
  1. How much do you currently crave opiates?
  2. In the past week, please rate how strong your desire to use opiates has been when something in the environment has reminded you of opiates?
  3. Please imagine yourself in the environment in which you previously used opiates. If you were in this environment today and if it were the time of day that you typically used opiates, what is the likelihood that you would use opiates today?
Short Opiate Withdrawal Scale-Gossop (SOWS-Gossop) | Weekly throughout Phase II (13 weeks)
  The SOWS-Gossop is an appropriate, precise, and sensitive measure to evaluate the symptoms of acute opioid withdrawal in research or clinical settings. The scale was derived from the original 32-item Opiate Withdrawal Scale to reduce redundancy while providing an equally sensitive measure of opioid withdrawal symptom severity appropriate for research and clinical practice. The assessment is a self-administered test used for the assessment of opiate withdrawal symptoms. The scale contains ten items: yawning, muscular tension, runny eyes, muscle twitching, pains, and aches, feeling of coldness, stomach cramps, insomnia, heart pounding, and feeling sick, making it easy and rapid to administer. The tool has a 4-point rating scale: 0 for 'none,' 1 for 'mild,' 2 for 'moderate,' and 3 for 'severe', with scores ranging from 0 to 30.
Proportion of patients who receive and tolerate an XR-NTX injection after acute detox treatment (Phase I) | One hour after receiving first XR-NTX injection (Phase II Day 1)

OTHER OUTCOMES:
Patient Health Questionnaire (PHQ-9) in Phase I | Baseline and Day 7
  The PHQ-9 is a validated tool in mental health and considered a powerful tool to assist clinicians with diagnosing depression and monitoring treatment response. The relationship between opioid use and depression is bidirectional. The PHQ-9 is a nine-item depression scale and is based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV. Each of the nine items is rated on a 0 (not at all) to 3 (nearly every day) scale. A total score is calculated by summing the nine items. Scores range from 0 to 27 and higher scores indicate a higher degree of depression.
Patient Health Questionnaire (PHQ-9) in Phase II | Monthly throughout Phase II (Day 28, 56, and 90)
  The PHQ-9 is a validated tool in mental health and considered a powerful tool to assist clinicians with diagnosing depression and monitoring treatment response. The relationship between opioid use and depression is bidirectional. The PHQ-9 is a nine-item depression scale and is based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV. Each of the nine items is rated on a 0 (not at all) to 3 (nearly every day) scale. A total score is calculated by summing the nine items. Scores range from 0 to 27 and higher scores indicate a higher degree of depression.
PTSD Checklist for DSM-5 (PCL-5) in Phase I | Baseline and Day 7
  Symptoms of post-traumatic stress disorder (PTSD) and opiate dependency may overlap, to which, opioid withdrawal symptoms may emulate PTSD hyperactive startle response. This is indicative a common physiological mechanism. The PCL-5 scale is the gold standard in PTSD assessment. It consisted of a 20-item self-report measurement that is capable of measuring symptom change during and after treatment. Additionally, the scale can provide a provisional PTSD diagnosis. Each of the 20 items is rated on a 0 (not at all) to 4 (extremely) scale. A total symptom severity score is calculated by summing the 20 items. Scores range from 0 and 80 and higher scores indicating a higher degree of PTSD symptomology. Evidence suggests that a10 to 20-point reduction in score represents a clinically significant change in PTSD symptoms.
PTSD Checklist for DSM-5 (PCL-5) in Phase II | Monthly throughout Phase II (Day 28, 56, and 90)
  Symptoms of post-traumatic stress disorder (PTSD) and opiate dependency may overlap, to which, opioid withdrawal symptoms may emulate PTSD hyperactive startle response. This is indicative a common physiological mechanism. The PCL-5 scale is the gold standard in PTSD assessment. It consisted of a 20-item self-report measurement that is capable of measuring symptom change during and after treatment. Additionally, the scale can provide a provisional PTSD diagnosis. Each of the 20 items is rated on a 0 (not at all) to 4 (extremely) scale. A total symptom severity score is calculated by summing the 20 items. Scores range from 0 and 80 and higher scores indicating a higher degree of PTSD symptomology. Evidence suggests that a10 to 20-point reduction in score represents a clinically significant change in PTSD symptoms.
Generalized Anxiety Disorder (GAD-7) in Phase I | Baseline and Day 7
  The GAD-7 is a valid and efficient tool for screening for GAD and assessing its severity in clinical practice and research. The questionnaire consists of 7 questions in which participants are asked to rate each item on a 0 (not at all) to 3 (nearly every day). GAD-7 total score for the seven items ranges from 0 to 21 where 0-4 represents minimal anxiety, 5-9 represents mild anxiety, 10-14 represents moderate anxiety and 15-21 represent severe anxiety.
Generalized Anxiety Disorder (GAD-7) in Phase II | Monthly throughout Phase II (Day 28, 56, and 90)
  The GAD-7 is a valid and efficient tool for screening for GAD and assessing its severity in clinical practice and research. The questionnaire consists of 7 questions in which participants are asked to rate each item on a 0 (not at all) to 3 (nearly every day). GAD-7 total score for the seven items ranges from 0 to 21 where 0-4 represents minimal anxiety, 5-9 represents mild anxiety, 10-14 represents moderate anxiety and 15-21 represent severe anxiety.
World Health Organization Quality of Life (WHOQOL-BREF) in Phase I | Baseline and Day 7
  The WHOQOL-BREF is a shorter version of the original assessment tool and is commonly used in clinical trials with participants undergoing substance use disorder intervention. The WHOQOL-BREF is comprised of 26-items and assesses the participant's quality of life across specific domains: physical health, psychological health, social relationships, and environment. In addition, there are 2 items that measure overall quality of life and general health. Participants rate how much they have experienced each item in the preceding 2 weeks on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely). Domain scores are scaled in a positive direction with higher scores denoting higher quality of life. The mean score of items within each domain is used to calculate the domain score. Raw domain scores will be converted to a 0 to 100 scale.
World Health Organization Quality of Life (WHOQOL-BREF) in Phase II | Monthly throughout Phase II (Day 28, 56, and 90)
  The WHOQOL-BREF is a shorter version of the original assessment tool and is commonly used in clinical trials with participants undergoing substance use disorder intervention. The WHOQOL-BREF is comprised of 26-items and assesses the participant's quality of life across specific domains: physical health, psychological health, social relationships, and environment. In addition, there are 2 items that measure overall quality of life and general health. Participants rate how much they have experienced each item in the preceding 2 weeks on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely). Domain scores are scaled in a positive direction with higher scores denoting higher quality of life. The mean score of items within each domain is used to calculate the domain score. Raw domain scores will be converted to a 0 to 100 scale.
Brief Assessment of Recovery Capital (BARC-10) from Phase I to Phase II | Baseline, Day 7, and monthly throughout Phase II (Day 28, 56, and 90)
  The BARC-10 is a short,10-item measure that examines recovery capital globally. Items were selected from the ARC for the BARC-10 using item response theory. The BARC-10 measures a unidimensional (i.e., global) construct of recovery capital across all the original 10 domains of the ARC. On average, it takes 2-5 minutes to complete. Scores range from 6-60. Individuals who have a recovery capital score of 47 or higher are likely to reach or sustain a year or longer of recovery from substance use disorder.
Short Opiate Withdrawal Scale-Gossop (SOWS-Gossop) in Phase II | Weekly throughout Phase II (13 weeks)
  The SOWS-Gossop is an appropriate, precise, and sensitive measure to evaluate the symptoms of acute opioid withdrawal in research or clinical settings. The scale was derived from the original 32-item Opiate Withdrawal Scale to reduce redundancy while providing an equally sensitive measure of opioid withdrawal symptom severity appropriate for research and clinical practice. The assessment is a self-administered test used for the assessment of opiate withdrawal symptoms. The scale contains ten items: yawning, muscular tension, runny eyes, muscle twitching, pains, and aches, feeling of coldness, stomach cramps, insomnia, heart pounding, and feeling sick, making it easy and rapid to administer. The tool has a 4-point rating scale: 0 for 'none,' 1 for 'mild,' 2 for 'moderate,' and 3 for 'severe', with scores ranging from 0 to 30.
14-Panel Urine Drug Screen in Phase I | Baseline and Day 7
  In Phase II, participants will provide a weekly urine sample to determine if opioids have been used in the past week (in conjunction with a self-report). A urine drug screen cup will be used to detect presence of: Amphetamines, Buprenorphine, Benzodiazepines, Cocaine, Ethyl Glucuronide, Fentanyl, Synthetic Marijuana, Ecstasy, Methamphetamines, Methadone, Opiates / Morphine, Oxycodone, Cannabinoid (Marijuana), and Tramadol. The urine drug screen cup also contains a temperature strip to confirm appropriate temperature of the sample and an adulteration panel for determination of sample tampering.
Xylazine Test Strip Screen in Phase I and Phase II | Baseline, Phase I Day 7, and weekly throughout Phase II (13 weeks)
  In addition to the 14-Panel Urine Drug Screen cup, a xylazine test strip will be used to detect the presence of xylazine in the urine.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Hazelden Betty Ford Foundation, Rancho Mirage, California
  - Gaudenzia, Inc., Crownsville, Maryland
  - Hazelden Betty Ford Foundation, Center City, Minnesota
  - Hazelden Betty Ford Foundation, Plymouth, Minnesota

DOCUMENTS (1):
  • Informed Consent Form (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT05053503/ICF_000.pdf